CLINICAL TRIAL: NCT03382301
Title: Impact of a Ciclosporin A Preconditioning for Prevention of Ischemia-reperfusion Injury After Renal Artery Stenosis Dilation
Brief Title: Ciclosporin A Preconditioning for Renal Artery Stenosis
Acronym: CicloSAAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 69HCL16_0823; 2017-002937-48 (EudraCT Number)
Record Dates: First submitted 2017-12-13; First posted 2017-12-22 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Renal Artery Stenosis
Keywords: Ischemia reperfusion injuries; Renal artery stenosis; Renal functional imaging
MeSH Terms: conditions — Renal Artery Obstruction; Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciclosporin A preconditioning (Experimental): Ciclosporin A preconditioning before renal artery stenosis dilation
  Interventions: Drug: Ciclosporin A preconditioning before renal artery stenosis dilation
- NaCl preconditioning (Placebo Comparator)
  Interventions: Drug: NaCl preconditioning before renal artery stenosis dilation

INTERVENTIONS:
Drug: Ciclosporin A preconditioning before renal artery stenosis dilation — Ciclosporin A perfusion (2.5 mg/kg) for 1 hour before renal artery dilation
  Arms: Ciclosporin A preconditioning
Drug: NaCl preconditioning before renal artery stenosis dilation — NaCl perfusion (Saline perfusion) for 1 hour (2.5 mg/kg) before renal artery dilation
  Arms: NaCl preconditioning

SUMMARY:
Renal artery stenosis is one the leading cause of secondary hypertension. Previous randomized controlled trials in humans have failed to demonstrate an improvement of renal function after stenosis dilation, probably because of a selection bias with more severe patients being excluded from randomization. Renal ischemia-reperfusion injuries have also not been taken into account. Indeed, reperfusion leads to a rapid renal blood flow recovery associated with renal ischemia-reperfusion injuries.

Mitochondrial permeability transition pore (mPTP) is a key player in the occurrence of ischemia reperfusion injuries because its opening leads to mitochondria leakage and cell death. However, preconditioning whether pharmacological or ischemic can prevent mPTP opening and protect cells. Ciclosporin A can prolong mPTP closing during reperfusion and reduce renal and cardiac tissular lesions. Another mPTP blocker (Bendavia) has been associated with an improvement of renal blood flow (RBF) and glomerular filtration rate (GFR) after renal artery stenosis dilation at 6 weeks in pigs. Based on a recent study, dilation overall benefit could be secondary to an improvement of the contralateral kidney GFR and tissue oxygen content, requiring a single kidney evaluation of those renal functional parameters. The investigators previously demonstrated that dose and timing of ciclosporin A preconditioning is key to protect kidneys from ischemia-reperfusion injuries. Previous controlled trials that failed to demonstrate a benefit of ciclosporin A conditioning have used post conditioning on necrotic cells. Considering kidney ischemia-reperfusion injuries, preconditioning have led to more encouraging results compared to ciclosporin A post conditioning in animals. Therefore the investigators aim to conduct the first clinical study of ciclosporin A preconditioning for prevention of kidney ischemia-reperfusion injuries after renal artery stenosis dilation.

Using renal functional imaging and the new PET-MRI (Positron Emission Tomography-Magnetic Resonance Imaging) combined device, the investigators will evaluate kidney perfusion, oxidative metabolism, glomerular filtration rate and oxygen content before and 3 months after renal artery stenosis dilation with or without a ciclosporin A preconditioning.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 50 years of age
* For women : only menopausal women
* Estimated Glomerular filtration rate ≥ 25 mL/min/1.73m2
* Renal artery stenosis with ≥ 70 % caliber reduction (Doppler or scanner or MRI)
* No controlateral stenosis
* Kidney size ≥ 7 cm
* Only atheromatous renal artery stenosis
* Resistant hypertension and/or rapid loss of kidney function and/or flash pulmonary edema
* Collective decision of dilation after a multidisciplinary meeting

Exclusion Criteria:

* Inclusion in another study
* Protected adults
* Person without a social security coverage
* Imprisoned person
* Systolic blood pressure >180 mmHg and/or diastolic blood pressure > 110 mmHg
* Non atheromatous renal artery stenosis
* Single kidney
* Multiple myeloma
* Iodine contrast agents allergy
* Ciclosporin A hypersensibility
* Severe other medical conditions that could be exacerbated by Iodine injection (cancer, lymphoma, active Hepatitis B, active Hepatitis C, uncontrolled HIV)
* Previous radiation exposure (above 20 mSv (millisievert) in the last 6 months before inclusion)
* MRI contra indications (MRI incompatible pacemaker or insulin pomp, metal clip, MRI incompatible cardiac valve, dental brace, claustrophobia)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Difference in relative increase (baseline and 3 months after) of global renal perfusion between the two groups | 3 months after renal artery stenosis dilation
  Global renal perfusion is assessed by 15O labeled water PET (Positron Emission Tomography) imaging

SECONDARY OUTCOMES:
Difference in the relative increase (baseline and 3 months after) of global renal oxidative metabolism between the two groups | 3 months after renal artery stenosis dilation
  Global renal oxidative metabolism is assessed by 11C labeled acetate PET (Positron Emission Tomography) imaging
Difference in the relative increase (baseline and 3 months after) of global renal oxygen content between the two groups | 3 months after renal artery stenosis dilation
  Global renal oxygen content is assessed by BOLD MRI (Blood-Oxygen-Level Dependent Magnetic Resonance Imaging)
Difference in the relative increase (baseline and 3 months after) of global glomerular filtration rate between the two groups | 3 months after renal artery stenosis dilation
  Global glomerular filtration rate is assessed by Iohexol measured clearance
Difference in the relative increase (baseline and 3 months after) of single-kidney perfusion (ischemic versus contralateral kidney) between the two groups | 3 months after renal artery stenosis dilation
  Kidney perfusion is assessed by 15O labeled water PET (Positron Emission Tomography) imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Exploration Fonctionnelle Rénale, Hôpital Edouard Herriot, Hospices Civils de Lyon, Lyon, France